CLINICAL TRIAL: NCT03000504
Title: A Randomized, Controlled Trial of the Use of a Dedicated Ballooned Intercostal Tube
Brief Title: Ballooned Intercostal Drain Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Royal Brompton & Harefield NHS Foundation Trust (Other)
Collaborators: Sherwood Forest Hospitals NHS Foundation Trust (Other); Oxford University Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 217496
Record Dates: First submitted 2016-11-25; First posted 2016-12-22 (Estimated); Last update posted 2018-05-16 (Actual); Status verified 2018-05

CONDITIONS: Pleural Effusion; Pneumothorax
MeSH Terms: conditions — Pleural Effusion; Pneumothorax

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ballooned intercostal drain (Experimental): Patients will have a Rocket Medical 16F ballooned chest drain inserted as per usual clinical guidelines. No other change to treatment will be made, and the drain is inserted in exactly the same way as a standard drain, using the Seldinger technique.
  Interventions: Device: Ballooned intercostal drain
- Standard intercostal drain (Active Comparator): Patients will have a standard 12F-16F Rocket Medical chest drain inserted as per usual clinical guidelines, using the Seldinger technique.
  Interventions: Device: Ballooned intercostal drain

INTERVENTIONS:
Device: Ballooned intercostal drain — Patients will have a Rocket Medical 16F ballooned intercostal drain inserted as per usual clinical guidelines. No other change to treatment will be made, and the drain is inserted in exactly the same way as a standard drain, using the Seldinger technique.

SUMMARY:
This study is designed to assess whether a new type of chest drain reduces the number of drains that fall out of or are accidentally removed from the chest cavity (usually requiring another drain to be inserted), without causing any increase in discomfort or other side-effects.

DETAILED DESCRIPTION:
Chest drains are an essential part of the treatment for patients with fluid or air around the lung, which usually causes breathlessness. Draining the fluid or air relieves symptoms and allows investigations to be carried out that can identify a cause for why the fluid or air is there. Chest drains are difficult to secure in place, and sometimes fall out despite the best possible care. This study tests a modified drain that has a small balloon near the end which, when inflated inside the chest cavity, should make it much harder for the drain to fall out of the chest. This was tested in a small pilot study, with encouraging results. The current study is comparing a group of patients treated with the new ballooned drain against a group treated with the standard drain, with patients equally but randomly allocated to each group. The chest drain has been through rigorous laboratory testing and has been CE marked for human use.

All patients requiring intercostal drainage for clinical reasons will be offered entry into the study, unless, in the view of the treating physician, blunt dissection is required. No other screening assessments will be required, other than the ability to sign the informed consent form.Patients who have provided signed informed consent will then proceed to the study protocol. Patients will be randomised to undergo either standard ICT insertion (usual clinical care) or insertion of the study drain using standard clinical policies and procedures at each participating centre.

Once a patient has been identified for the trial and has signed the informed consent form, baseline details will be entered into a dedicated web-based programme accessible at all sites, and patients will be allocated 1:1 to either usual care or to the study drain.

All subsequent care will be as per best clinical care for all patients in both arms of the study. The only additional assessments over and above usual care will be the collection of pain scores. Pain will be rated by the patients on a visual analogue scale (VAS) on up to 4 occasions - insertion, 24 and 72 hours post insertion, and at drain removal.

ELIGIBILITY:
Inclusion Criteria:

1. Age >16 years
2. Able to give written informed consent
3. Requiring intercostal tube drainage for clinical reasons

Exclusion Criteria:

1. Inability to provide written informed consent
2. Requiring blunt dissection for intercostal tube insertion
3. Haemothorax

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Estimated)
Dates: Start 2018-03-07 (Actual); Primary Completion 2019-06 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
The difference in the percentage of accidental removal of ICTs between study arms | Up to 1 week dependent upon duration of intercostal drainage
  The number of drains prematurely and unintentionally removed from the pleural space

SECONDARY OUTCOMES:
The difference in patient reported pain scores, using a visual analogue scale | At drain insertion, 24hrs post-insertion, 72hrs-post insertion, and at drain removal, usually a maximum of 7 days
The frequency of balloon rupture | Up to 1 week dependent upon duration of intercostal drainage
The difference in duration of drainage between the study arms | Up to 1 week dependent upon duration of intercostal drainage
Cost-effectiveness profiles for each intervention | Up to 1 week dependent upon duration of intercostal drainage

CONTACTS AND LOCATIONS:
Overall Officials: Samuel V Kemp, MBBS, MD, Principal Investigator — Royal Brompton and Harefield NHS Foundation Trust
Locations (3):
- United Kingdom (3):
  - Sherwood Forest Hospitals NHS Foundation Trusty, Sutton in Ashfield, Nottinghamshire
  - Oxford Respiratory Trials Unit, Oxford, Oxfordshire
  - Royal Brompton Hospital, London

IPD SHARING:
Plan to Share IPD: No